CLINICAL TRIAL: NCT00041574
Title: Development of a Hospital-Based Home Program for the Use of Inhaled Nitric Oxide in the Chronic Management of Severe Cardiopulmonary Diseases
Brief Title: Hospital-Based Program for Treatment of Severe Cardiopulmonary Disease With Inhaled Nitric Oxide
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed for lack of enrollment
Sponsor: Mallinckrodt (Industry)
Responsible Party: Robert Small, INO Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INOT-31
Record Dates: First submitted 2002-07-10; First posted 2002-07-11 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Hypertension; Lung Disease; Sickle Cell Disease; Cardiac Transplant; Lung Transplant
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases; Anemia, Sickle Cell | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Inhaled Nitric Oxide will be delivered through the INOpulse® at a Low Dose Range (3mL to 10mL; in 1mL increments) and Ultra Low Dose Ranges (0.5mL to 4mL; 0.5mL, then 1 to 4mL in 1mL increments).
  Interventions: Drug: Inhaled Nitric Oxide

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Inhaled Nitric Oxide will be delivered through the INOpulse® at a Low Dose Range (3mL to 10mL; in 1mL increments) and Ultra Low Dose Ranges (0.5mL to 4mL; 0.5mL, then 1 to 4mL in 1mL increments).
  Other Names: INOmax®

SUMMARY:
The purpose of this program is to evaluate the logistic issues and patient requirements for chronic pulsed INOmax delivery in ambulatory, home-care patients. To understand patient needs, patients with a variety of underlying diseases will be included. Safety of chronic therapy will be monitored by serial measurements of methemoglobin, platelet function assay and reported adverse events.

DETAILED DESCRIPTION:
This study will help develop a comprehensive home care program using INOmax delivery systems. This study will enroll a limited number of patients (5-7) from several disease categories in order to develop the experience with testing acute and chronic responsiveness to INO therapy. The following groups will be tested:

1. Primary pulmonary hypertension (PPH)
2. Severe pulmonary hypertension due to congenital (anatomic) heart disease
3. Pulmonary hypertension or severe impairment of gas exchange in infants and children with chronic lung disease
4. Pulmonary hypertension or severe impairment of gas exchange due to severe chronic lung disease in adults
5. Pulmonary hypertension or severe impairment of gas exchange in hematologic and transplant disorders - young children and adults with sickle cell disease, chronic lung disease after bone marrow transplant, cardiac transplant, or lung transplant

ELIGIBILITY:
Inclusion criteria:

* Patients with pulmonary arterial hypertension (PAH) as defines by a mean pulmonary artery pressure (PAP) of 25 mmHg or greater by cardiac catheterization within the previous 12 months AND/OR Patients with chronic lung disease with severe impairment of gas exchange unresponsive to conventional medical management.
* If patient is receiving prostacyclin infusion treatment it must have been started at least one month prior to starting INO therapy. Patients will not be withdrawn from the study if started on other medications for treatment of pulmonary hypertension.
* Ability to establish a clinical investigator and a drug shipment site in the local area.

Exclusion Criteria:

* The Principal Investigator has determined that the patient and/or caregiver is/are unable to manage safe administration of home nitric oxide therapy and maintain appropriate drug accountability and storage.
* Women who are pregnant or nursing.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Methemoglobin level | 24 and 72 hours after treatment start, then at 1, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Vital Signs | taken at 1, 2, 3, 4, 24, and 72 hours after treatment begins, then at 1, 3, 6, 9 and 12 months
Pulse Oximetry | taken at 1, 2, 3, 4, 24, and 72 hours after treatment start and then at 1, 3, 6, 9 and 12 months
Adverse Event Occurence | Study Duration
Echocardiogram | At 72 hours after treatment start, then at 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Abman, MD, Principal Investigator — Children's Hospital Colorado
Locations (3):
- United States (3):
  - The Children's Hospital, Denver, Colorado
  - University of Colorado Hospital, Denver, Colorado
  - Rhode Island Hospital, Providence, Rhode Island